CLINICAL TRIAL: NCT06688643
Title: The Impact of Intrathecal Morphine Versus Continuous Epidural Analgesia on Return of Bowel Function in Patients Undergoing Laparoscopic Ileal Conduit : a Prospective, Randomized Controlled Trial
Brief Title: The Impact of Intrathecal Morphine Versus Continuous Epidural Analgesia on Return of Bowel Function in Patients Undergoing Laparoscopic Ileal Conduit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaguang Duan (Other)
Responsible Party: Sponsor-Investigator, Xiaguang Duan, Deputy Chief of Anesthesiology, Inner Mongolia Baogang Hospital
Organization: Inner Mongolia Baogang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-MER-206
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2021-10

CONDITIONS: Bladder Cancer
Keywords: Bowel function; Continuous epidural analgesia (CEA); intrathecal morphine(ITM); laparoscopic ileal conduit (Bricker); Postoperative nausea and vomiting(PONV); Pruritus
MeSH Terms: conditions — Urinary Bladder Neoplasms; Postoperative Nausea and Vomiting; Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ITM group (Experimental): Patients in the ITM group underwent intrathecal injection with 0.2 mg morphine after admission to the operating room.
  Interventions: Device: ITM group
- EA group (Experimental): Patients in the EA group underwent epidural anesthesia after admission to the operating room. Following successful epidural puncture, 3 ml of 2% lidocaine was administered. Once the block level was confirmed, the epidural analgesia pump was activated, delivering 8 ml/h of 0.1% ropivacaine.
  Interventions: Device: EA group

INTERVENTIONS:
Device: ITM group — Patients in the ITM group underwent intrathecal injection with 0.2 mg morphine after admission to the operating room.Mechanical ventilation was initiated in pressure-regulated volume control (PRVC) mode after induction. Ventilator settings (Aestiva; GE Healthcare, Waukesha, Wisconsin, USA) were as follows: tidal volume 6-8 ml kg-1, positive end-expiratory pressure (PEEP) 0 cmH2O, inspiratory-to-expiratory ratio 1:2, respiratory rate 16 beats per minute (BPM), and inspired oxygen concentration 41%.
  Arms: ITM group
Device: EA group — Patients in the EA group underwent epidural anesthesia after admission to the operating room. Following successful epidural puncture, 3 ml of 2% lidocaine was administered. Once the block level was confirmed, the epidural analgesia pump was activated, delivering 8 ml/h of 0.1% ropivacaine.Mechanical ventilation was initiated in pressure-regulated volume control (PRVC) mode after induction. Ventilator settings (Aestiva; GE Healthcare, Waukesha, Wisconsin, USA) were as follows: tidal volume 6-8 ml kg-1, positive end-expiratory pressure (PEEP) 0 cmH2O, inspiratory-to-expiratory ratio 1:2, respiratory rate 16 beats per minute (BPM), and inspired oxygen concentration 41%.
  Arms: EA group

SUMMARY:
This study aims to compare the effects of intrathecal morphine (ITM) and continuous epidural analgesia (CEA) on bowel function recovery after Bricker surgery.This study was a prospective, randomized controlled trial that included 72 patients with bladder cancer undergoing elective Bricker surgery, who were randomly assigned to either the ITM group (n=36) or the CEA group (n=36). Postoperatively, patients in both groups received either ITM or CEA for pain management, and postoperative bowel function recovery time, pain scores, PONV, itching, and other indicators were recorded.

DETAILED DESCRIPTION:
Patients This study was approved by the Medical Ethics Committee of Baogang Hospital, Inner Mongolia (2021-MER-206) on October 11, 2021, and adhered to the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) guidelines. All participants provided informed consent voluntarily. From January 25, 2022, to November 1, 2024, 72 patients (aged 50-90 years) with bladder cancer undergoing elective Bricker surgery were enrolled at Baogang Hospital, Inner Mongolia. All patients were classified as ASA I-III. Patients were excluded if they had allergies to any anesthetic agents used in this study or if they had adverse reactions to any of the analgesics included in the study. Patients who refused to sign the consent form or were uncooperative were deemed ineligible for clinical evaluation. Patients were excluded if they had uncontrolled hypertension, hypersensitivity to pain, a history of gastrointestinal disease, impaired cardiopulmonary function, cerebrovascular disease, sleep disorders, or psychiatric disorders.

Randomization and blinding Patients were randomly assigned to the ITM group (n=36) or EA group (n=36) using a random number table. Patients in the ITM group underwent intrathecal injection with 0.2 mg morphine after admission to the operating room. Patients in the EA group underwent epidural anesthesia after admission to the operating room. Following successful epidural puncture, 3 ml of 2% lidocaine was administered. Once the block level was confirmed, the epidural analgesia pump was activated, delivering 8 ml/h of 0.1% ropivacaine. General anesthesia with endotracheal intubation was administered to both groups after the aforementioned procedures. Patients and surgeons were blinded to group assignment, while the anesthesiologists and nurses administering anesthesia were aware of the group allocation.

General anesthesia and monitoring Upon arrival in the operating room, patients were monitored for pulse oximetry (SPO2), electrocardiogram (ECG), bispectral index (BIS), and non-invasive arterial blood pressure. Pain threshold (PTh, mA) and pain tolerance threshold (PTTh, mA) were measured and recorded. Patients received pre-operative administration of Penehyclidine Hydrochloride Injection (Lot H20051948, Chengdu List Pharmaceutical Co., Ltd., China) (0.01 mg kg-1 i.v.). Induction was achieved with propofol (1.5-2 mg kg-1 i.v.), rocuronium bromide (1-2 mg kg-1 i.v.), and fentanyl (1-2 μg kg-1 i.v.). Anesthesia was maintained with inhaled sevoflurane or desflurane, with the inhaled concentration adjusted according to BIS values. Remifentanil (0.05-0.2 μg kg-1 min-1 i.v.) was continuously infused to maintain blood pressure and heart rate within ±20% of baseline values. Mechanical ventilation was initiated in pressure-regulated volume control (PRVC) mode after induction. Ventilator settings (Aestiva; GE Healthcare, Waukesha, Wisconsin, USA) were as follows: tidal volume 6-8 ml kg-1, positive end-expiratory pressure (PEEP) 0 cmH2O, inspiratory-to-expiratory ratio 1:2, respiratory rate 16 beats per minute (BPM), and inspired oxygen concentration 41%. The patient was positioned in the Trendelenburg position, with the operating table tilted 20-25° head down. Carbon dioxide pneumoperitoneum was established at an intra-abdominal pressure of 10-15 mmHg.

Postoperative care Vital signs were monitored in the Post Anesthesia Care Unit (PACU), with supplemental oxygen provided via facemask. For hypotension, ephedrine (6-10 mg) was administered, and fluid administration was increased. Atropine (0.3-0.5 mg) was given for bradycardia. For pain, sufentanil (0.1-0.2 μg/kg) was administered.

Data collection Upon arrival in the operating room, HR (bpm), mean arterial pressure (MAP, mmHg) (calculated as MAP = diastolic pressure + 1/3 pulse pressure), BIS, remifentanil dosage (mg), ephedrine dosage (mg), duration of surgery (minutes), and duration of anesthesia (minutes) were recorded for all patients.

In the PACU, the following data were recorded: number of patients requiring sufentanil (μg), number of patients experiencing respiratory depression (n), number of hypotension events requiring intervention (n), ephedrine dosage (mg), intravenous fluid volume (ml), number of patients experiencing bradycardia (n), atropine dosage (mg), Bromage score, and time spent in the PACU (min). For patients transferred to the high dependency unit, the number of patients (n) and length of stay (h) were recorded.

Postoperatively, rest pain (Numerical Rating Scale, NRS), dynamic pain (NRS), morphine equivalent (mg), quality of sleep on the first night (Likert scale, 1-5), functional recovery (return of bowel function, h, recommencement of oral intake, h, and time to first mobilization, h), quality of recovery (QoR, 0-15) on postoperative day 1, and hospital stay (days) were recorded at 4, 8, 12, and 24 hours. Ketorolac dosage (mg), hydromorphone dosage (mg), oral medications, number of episodes of PONV (n), antiemetic dosage (mg), number of episodes of pruritus (n), and Comprehensive Complication Index (CCI) were recorded over 24 hours.

Statistical analysis Sample size estimation was conducted using PASS 21.0.3 software (NCSS, LLC, Kaysville, Utah, USA), selecting the "Two-Sample T-Tests Allowing Unequal Variance" module10,11. With sample sizes of 23 in each group, a two-sided, two-sample t-test with unequal variances achieves 91.25% power to reject the null hypothesis of equal means at a significance level (alpha) of 0.05.The calculated results indicated an average group sample size (n) of 23, a 20% dropout rate, and a dropout-inflated expected enrollment sample size of 29.

Data were presented as means (standard deviations), frequencies (%), or medians (Confidence Interval). All statistical analyses were conducted using GraphPad Prism software version 10.2.3. The Kolmogorov-Smirnov test was performed to investigate the normality of the distribution of continuous variables. An independent t test or Mann-Whitney U test was performed to compare continuous variables, as appropriate. The x2 test or Fisher's exact was performed to compare categorical variables. Repeated-measures analysis of variance was performed to compare changes in some variables over time. Statistical significance was set at P value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* All participants provided informed consent voluntarily
* ASA I-III

Exclusion Criteria:

* allergies to any anesthetic agents used in this study
* refused to sign the consent form
* uncooperative were deemed ineligible for clinical evaluation
* hypersensitivity to pain
* a history of gastrointestinal disease
* sleep disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
bowel function recovery time | 24 hours after surgery
  12 hours indicates good bowel function, 24 hours indicates good bowel function.

SECONDARY OUTCOMES:
pain scores | 24 hours after surgery
  Zero is equivalent to no pain and 10 indicates the worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: January 2025-January 2026
Access Criteria: Anyone needing IPD information, contact the author at email: alonlord2023@gmail.com